CLINICAL TRIAL: NCT00879255
Title: Telemental Health and Cognitive Processing Therapy for Rural Combat Veterans With PTSD
Brief Title: Telemental Health and Cognitive Processing Therapy for Rural Combat Veterans With Posttraumatic Stress Disorder
Acronym: CPTVTEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHI 07-259; 2008-05_LM_Promise 0005 (Other: VAPHICS IRB); PT074516 (Other Grant/Funding Number: CDMRP); NCT00769977 (obsolete NCT alias)
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: cognitive processing therapy; combat; veterans; PTSD; Telemental Health; Videoteleconference; outcome; Rural; Remote; CPT; VTC
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videoteleconferencing CPT (Experimental): The experimental arm is the group condition that received the CPT treatment via videoteleconferencing modality as compared to the experimental condition which is via face-to-face traditional modality.
  Cognitive Processing Therapy Group Videoteleconference is delivered to male combat veterans who have been diagnosed with PTSD, through videoteleconference.
  Interventions: Behavioral: Cognitive Processing Therapy Group Videoteleconference
- Face-to-Face CPT (Active Comparator): The control arm is the group condition that received the CPT treatment via face-to-face traditional modality as compared to the experimental condition which is via videoteleconferencing modality.
  Cognitive Processing Therapy Group In-Person is delivered to male combat veterans who have been diagnosed with PTSD, in-person, rather than through videoteleconference.
  Interventions: Behavioral: Cognitive Processing Therapy Group In-Person

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy Group Videoteleconference — Cognitive Processing Group Therapy is delivered to male combat veterans who have been diagnosed with PTSD, through videoteleconference.
  Other Names: CPT-VT
  Arms: Videoteleconferencing CPT
Behavioral: Cognitive Processing Therapy Group In-Person — Cognitive Processing Group Therapy is delivered to male combat veterans who have been diagnosed with PTSD, in-person, rather than through videoteleconference.
  Other Names: CPT-NP
  Arms: Face-to-Face CPT

SUMMARY:
The immediate objective of this project was to evaluate the clinical effectiveness of a telemental health modality (video-teleconferencing) for providing an evidence-based group intervention (Cognitive Processing Therapy; CPT) to rural OIF/OEF Reservists, National Guardsmen, and veterans suffering with PTSD.

DETAILED DESCRIPTION:
The project was a 5-year prospective randomized clinical trial which conducted a direct comparison of the VTC and in-person modalities using rigorous methodology and a sophisticated analysis of equivalency between clinical and process outcome domains. In addition, cost effectiveness of this modality will be addressed. Approximately 130 combat Reservists, National Guardsmen, or veterans were recruited from multiple clinical sites. Prospective participants received a comprehensive assessment at baseline to determine eligibility. The exclusion criteria selected are consistent with large PTSD randomized clinical trials as well as research using the CPT protocol with military populations with PTSD. The treatment was delivered twice a week over 6 weeks by a doctoral level psychologist. Quality control procedures were incorporated into the study's design to ensure integrity, fidelity and standard administration of the CPT intervention across both conditions. Participants received additional assessments at mid-treatment, immediately post-treatment, and at 3 and 6 months post-treatment. Outcome domains include: 1) clinical outcomes (symptom severity, social functioning); 2) process outcomes (perception of treatment, satisfaction, group therapy alliance, treatment compliance, and attrition and treatment credibility); and (3) cost-effectiveness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of current combat related PTSD determined by the Clinician Administered PSTD Scale (CAPS-IV)
* participants taking psychoactive medications have to have a stable regimen for at least 45 days prior to study entry

Exclusion Criteria:

* active psychotic symptoms/disorder as determined by the SCID for DSM-IV
* active homicidal or suicidal ideation as determined by the structured clinical interview
* any significant cognitive impairment or history of Organic Mental Disorder as determined by the structured clinical interview
* active (current) substance dependence as determined by the SCID (lifetime substance dependence/abuse not excluded)
* unwillingness to refrain from substance abuse during treatment
* female veterans

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-10; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Morland, PsyD, Principal Investigator — VA Pacific Islands Health Care System, Honolulu, HI
Locations (1):
- VA Pacific Islands Health Care System, Honolulu, HI, Honolulu, Hawaii, United States

REFERENCES:
- [Result] Morland LA, Greene CJ, Rosen C, Mauldin PD, Frueh BC. Issues in the design of a randomized noninferiority clinical trial of telemental health psychotherapy for rural combat veterans with PTSD. Contemp Clin Trials. 2009 Nov;30(6):513-22. doi: 10.1016/j.cct.2009.06.006. Epub 2009 Jul 1. PMID 19576299
- [Result] Morland LA, Hynes AK, Mackintosh MA, Resick PA, Chard KM. Group cognitive processing therapy delivered to veterans via telehealth: a pilot cohort. J Trauma Stress. 2011 Aug;24(4):465-9. doi: 10.1002/jts.20661. Epub 2011 Jul 25. PMID 21793047
- [Result] Morland LA, Mackintosh MA, Greene CJ, Rosen CS, Chard KM, Resick P, Frueh BC. Cognitive processing therapy for posttraumatic stress disorder delivered to rural veterans via telemental health: a randomized noninferiority clinical trial. J Clin Psychiatry. 2014 May;75(5):470-6. doi: 10.4088/JCP.13m08842. PMID 24922484
- [Derived] Glassman LH, Mackintosh MA, Wells SY, Wickramasinghe I, Walter KH, Morland LA. Predictors of Quality of Life Following Cognitive Processing Therapy Among Women and Men With Post-Traumatic Stress Disorder. Mil Med. 2020 Jun 8;185(5-6):e579-e585. doi: 10.1093/milmed/usz474. PMID 32077948
- [Derived] Raab PA, Mackintosh MA, Gros DF, Morland LA. Examination of the Content Specificity of Posttraumatic Cognitions in Combat Veterans With Posttraumatic Stress Disorder. Psychiatry. 2015;78(4):328-40. doi: 10.1080/00332747.2015.1082337. PMID 26745686
- [Derived] Raab PA, Mackintosh MA, Gros DF, Morland LA. Impact of comorbid depression on quality of life in male combat Veterans with posttraumatic stress disorder. J Rehabil Res Dev. 2015;52(5):563-76. doi: 10.1682/JRRD.2014.05.0130. PMID 26466310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included 13 group cohorts plus 1 pilot group cohort. Not counting the cohort 1 pilot, approximately 246 combat Reservists, National Guardsmen, or Veterans from multiple VA Pacific Island Health Care System clinical sites were assessed for eligibility, and 125 were subsequently randomized into treatment groups.
Pre-assignment Details: Not counting the cohort 1 pilot group, approximately 246 combat Reservists, National Guardsmen, or Veterans received a comprehensive assessment at baseline to determine eligibility. 144 met inclusion criteria, 19 declined participation, for 125 ITT who were randomized into treatment groups.
Groups:
- Videoteleconferencing CPT: The experimental arm is the group condition that received the CPT treatment via videoteleconferencing modality as compared to the experimental condition which is via face-to-face traditional modality.
  Cognitive Processing Therapy Group Videoteleconference is delivered to male combat veterans who have been diagnosed with PTSD, through videoteleconference.
  Cognitive Processing Therapy Group Videoteleconference: Cognitive Processing Group Therapy is delivered to male combat veterans who have been diagnosed with PTSD, through videoteleconference.
- Face-to-Face CPT: The control arm is the group condition that received the CPT treatment via face-to-face traditional modality as compared to the experimental condition which is via videoteleconferencing modality.
  Cognitive Processing Therapy Group In-Person is delivered to male combat veterans who have been diagnosed with PTSD, in-person, rather than through videoteleconference.
  Cognitive Processing Therapy Group In-Person: Cognitive Processing Group Therapy is delivered to male combat veterans who have been diagnosed with PTSD, in-person, rather than through videoteleconference.
Period: Overall Study
Arm/Group | Videoteleconferencing CPT | Face-to-Face CPT
Started | 61 | 64
Received Allocated Intervention: | 51 | 56
Completed Posttreatment Follow-up | 50 | 55
Completed 3-mo Follow-up | 48 | 49
Completed | 45 (Completed 6-mo follow-up) | 45 (Completed 6-mo follow-up)
Not Completed | 16 | 19

BASELINE CHARACTERISTICS:
Population: Male combat veterans with posttraumatic stress disorder (PTSD).
Groups:
- Total: Total of all reporting groups
Arm/Group | Videoteleconferencing CPT | Face-to-Face CPT | Total
Number analyzed (Participants) | 61 | 64 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (11.8) | 54.6 (13.2) | 55.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 64 | 125
Region of Enrollment [Number; unit: participants]
  United States | 61 | 64 | 125

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale, for DSM-IV (CAPS IV)
Description: The CAPS is a 30-item interview measure that assesses the frequency and intensity of PTSD symptoms during the past month and the impact these symptoms have had on social and occupational functioning. The CAPS also provides a global scale score of PTSD severity (range 0 - 136) with higher scores indicating worse symptoms, which was used as the primary outcome measure. Scores reported here are differences between individuals follow up scores (e.g. post-treatment CAPS score assessed at two-weeks following end of treatment) minus their baseline CAPS scores, such that negative numbers represent reductions in CAPS scores (or improvement) over time.
Time Frame: Post-treatment (two-weeks following end of treatment)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Videoteleconferencing CPT | Face-to-Face CPT
Number analyzed (Participants) | 61 | 64
units on a scale | -15.97 (3.21) | -11.22 (2.89)
Statistical Analysis 1: Comparison: Videoteleconferencing CPT vs Face-to-Face CPT; Test type: Non-Inferiority or Equivalence — We used a noninferiority design to test the hypothesis that VTC is noninferior to in-person treatment delivery. The noninferiority margin was determined to be 10 CAPS points. We analyzed means differences in CAPS scores between the two treatment conditions (VTC minus in-person) with positive values indicating greater reductions in VTC condition. Power was estimated to be 90% with alpha = .20, and a between-group difference equaling an effect size of d = .50 (estimated 10 CAPS points); p > .05, noninferiority analysis — The noninferiority margin is the maximum clinically meaningful amount by which VTC can be "worse than" the in-person delivery to allow for a conclusion of noninferiority (a priori set to 10 CAPS points); We hypothesized that VTC is noninferior to in-person condition, which is supported if upper limit of 95% CI is less than preset noninferiority margin; Mean Difference (Final Values) = -4.75, 95% CI 2-sided [-11.92 to 2.42] — The noninferiority hypothesis would be supported if the 95% Confidence Interval of the difference in CAPS scores between the 2 conditions (VTC minus in-person scores) is less than the present noninferiority margin (10 CAPS points)

2. Primary Outcome: Clinician Administered PTSD Scale, for DSM-IV (CAPS IV)
Description: The CAPS is a 30-item interview measure that assesses the frequency and intensity of PTSD symptoms during the past month and the impact these symptoms have had on social and occupational functioning. The CAPS also provides a global scale score of PTSD severity (range 0 - 136) with higher scores indicating worse symptoms, which was used as the primary outcome measure. Scores reported here are differences between individuals follow up scores (e.g. 3-month post-treatment) minus their baseline CAPS scores, such that negative numbers represent reductions in CAPS scores (or improvement) over time.
Time Frame: 3-month Post-treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Videoteleconferencing CPT | Face-to-Face CPT
Number analyzed (Participants) | 61 | 64
units on a scale | -14.22 (3.72) | -9.46 (3.32)
Statistical Analysis 1: Comparison: Videoteleconferencing CPT vs Face-to-Face CPT; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, noninferiority design — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.76, 95% CI 2-sided [-11.65 to 2.13] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Clinician Administered PTSD Scale, for DSM-IV (CAPS IV)
Description: The CAPS is a 30-item interview measure that assesses the frequency and intensity of PTSD symptoms during the past month and the impact these symptoms have had on social and occupational functioning. The CAPS also provides a global scale score of PTSD severity (range 0 - 136) with higher scores indicating worse symptoms, which was used as the primary outcome measure. Scores reported here are differences between individuals follow up scores (e.g. 6-month post-treatment) minus their baseline CAPS scores, such that negative numbers represent reductions in CAPS scores (or improve) over time.
Time Frame: 6 months post-treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Videoteleconferencing CPT | Face-to-Face CPT
Number analyzed (Participants) | 61 | 64
units on a scale | -15.17 (3.52) | -9.61 (3.29)
Statistical Analysis 1: Comparison: Videoteleconferencing CPT vs Face-to-Face CPT; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > .05, noninferiority test — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.56, 95% CI 2-sided [-16.26 to 5.14] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: The study was monitored for adverse events from 2009 to 2013.
Description: At the onset of study a committee was established among the investigators that guided protocol monitoring of any unanticipated problems involving risk to participants or others (UPRs) (which includes serious adverse events) that could occur in the study.
Arm/Group | Videoteleconferencing CPT | Face-to-Face CPT
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/64
Other Adverse Events (participants affected / at risk) | 0/61 | 0/64

LIMITATIONS AND CAVEATS:
For patients in rural areas, their local mental health facilities may not have access to videoteleconferencing technology.There were no women veterans as study participants. Participants with acute safety concerns or current substances were excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No